CLINICAL TRIAL: NCT04239157
Title: A Phase II, Open-Label, Study of Subcutaneous Canakinumab, an Anti-IL-1β Human Monoclonal Antibody, for Patients With Low or Int-1 Risk IPSS/IPSS-R Myelodysplastic Syndromes and Chronic Myelomonocytic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0339; NCI-2019-08494 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0339 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-12-31; First posted 2020-01-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome; Recurrent Chronic Myelomonocytic Leukemia; Recurrent Myelodysplastic Syndrome; Refractory Chronic Myelomonocytic Leukemia; Refractory Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (canakinumab) (Experimental): Patients receive canakinumab SC on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Canakinumab

INTERVENTIONS:
Biological: Canakinumab — Given SC
  Other Names: ACZ885; Ilaris

SUMMARY:
This phase II trial studies how well canakinumab works for the treatment of low- or intermediate-risk myelodysplastic syndrome or chronic myelomonocytic leukemia. Canakinumab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

- To assess the clinical activity of canakinumab in patients with low or intermediate-1 myelodysplastic syndrome (MDS) or CCUS.

SECONDARY OBJECTIVES:

* To assess the safety profile of canakinumab in patients with low or intermediate-1 risk by - IPSS or IPSS-R score ≤3.5 MDS, CCUS
* To assess the rate of transfusion independence (TI)
* To assess duration of response

EXPLORATORY OBJECTIVE:

- To assess pharmacodynamic (PD) parameters of canakinumab

OUTLINE:

Patients receive canakinumab subcutaneously (SC) on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years as MDS and CCUS are very rare conditions in the pediatric setting.
* Cohorts 1-3: Diagnosis of MDS according to WHO 2016 classification and low or intermediate-1 risk by IPSS or IPSS-R with a score of ≤ 3.5.
* Cohort 4: Diagnosis of CCUS defined as:
* Presence of a somatic pathogenic variant associated with hematological malignancy without morphological evidence of myelodysplasia
* Variant allele fraction of greater than or equal to 2% in at least one identified somatic pathogenic variant
* Bone marrow aspirate excluding hematological malignancy and MDS

  * Presence of a cytopenia for >30 days. Cytopenia will be defined using accepted CHRS (Clonal Hematopoiesis Risk Score) criteria (Weeks et al, NEJM Evidence in press): ANC <1.8 or hgb <12 in females and <13 in males or a platelet count of <150.
* Cohort 1: Participants need to have not responded to prior therapy with ESAs or hypomethylating agents (HMAs). These could include azacitidine, decitabine, SGI-110, ASTX727, or CC-486. Patients will need to have received at least 4 cycles of HMA. Participants with relapse or progression after any number of cycles of HMA by IWG 2006 criteria will also be candidates. Participants with evidence of del 5q alteration also are required to have been treated with Lenalidomide.
* Cohort 1: Hemoglobin <10g/dL with symptomatic anemia or transfusion dependency defined as the need for prior transfusion in the past 8 weeks for a hemoglobin level less than 8g/dl.
* Cohort 2: Transfusion dependency defined as the need for prior transfusion in the past 8 weeks of (1) at least 2 units of PRBC for a hemoglobin level less than 8g/dl or symptomatic anemia (hemoglobin <10g/dL), or (2) any platelet transfusion.
* Participants (or patient's legally authorized representative) must have signed an informed consent document indicating that the patient understands the purpose of and procedures required for the study and is willing to participate in the study.
* Adequate hepatic function with total bilirubin </=3 x ULN, AST or ALT </= 3xULN.
* Serum creatinine clearance >30mL/min and no end/stage renal disease (using Cockcroft-Gault).
* ECOG performance status </=2.

Exclusion Criteria:

* Active infection not adequately responding to appropriate antibiotics.
* Prior treatment with IL-1/IL-1r inhibitors
* Absolute neutrophil count (ANC) <0.5x109 k/ul; colony-stimulating factors can be administered prior to study drug initiation.
* Female participants who are pregnant or lactating.
* Participants with reproductive potential who are unwilling to following contraception requirements (including condom use for males with sexual partners, and for females: prescription oral contraceptives [birth control pills], contraceptive injections, intrauterine devices [IUD], double-barrier method [spermicidal jelly or foam with condoms or diaphragm], contraceptive patch, or surgical sterilization) throughout the study. Reproductive potential is defined as no previous surgical sterilization or females that are not post-menopausal for 12 months.
* Female participants with reproductive potential who do not have a negative urine or blood beta-human chorionic gonadotropin (beta HCG) pregnancy test at screening.
* History of an active malignancy within the past 2 years prior to study entry, with the exception of: a. Adequately treated in situ carcinoma of the cervix uteri b. Adequately treated basal cell carcinoma or localized squamous cell carcinoma of the skin or any other malignancy with a life expectancy of more than 2 years.
* Participants receiving any other concurrent investigational agent or chemotherapy, radiotherapy, or immunotherapy (within 14 days of initiating study treatment).
* Known history of testing positive for Human Immunodeficiency Virus (HIV) infections.

Participants requiring systemic steroids, methotrexate or other immunosuppressive drugs will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hematological improvement (HI) | After 2 cycles (each cycle is 28 days)
  Will be monitored simultaneously using the Bayesian approach of Thall, Simon, Estey. Will estimate the HI rate for canakinumab, along with the 95% credible intervals. The association between HI rate and patient's clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test.
Incidence of adverse events | Up to 4 weeks
  Will be monitored simultaneously using the Bayesian approach of Thall, Simon, Estey. Safety data of the patients will be summarized using descriptive statistics such as mean, standard deviation, median and range. Toxicity type, severity and attribution will be summarized for each patient using frequency tables.

SECONDARY OUTCOMES:
Transfusion independence | Up to 2 years
Duration of response | Up to 2 years
  Will be summarized using descriptive statistics such as mean, standard deviation, median and range.
Progression-free survival (PFS) | Up to 2 years
  Will be estimated using the method of Kaplan and Meier. Comparisons of time-to-time event endpoints by important subgroups will be made using the log-rank tests.
Leukemia-free survival (LFS) | Up to 2 years
  Will be estimated using the method of Kaplan and Meier. Comparisons of time-to-time event endpoints by important subgroups will be made using the log-rank tests.
Overall survival (OS) | Up to 2 years
  Will be estimated using the method of Kaplan and Meier. Comparisons of time-to-time event endpoints by important subgroups will be made using the log-rank tests.

OTHER OUTCOMES:
Pharmacodynamic (PD) parameters of canakinumab | Up to 2 years
  Will include Correlative studies.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Rodriguez-Sevilla JJ, Adema V, Chien KS, Loghavi S, Ma F, Yang H, Montalban-Bravo G, Huang X, Calvo X, Joseph J, Bodden K, Garcia-Manero G, Colla S. The IL-1beta inhibitor canakinumab in previously treated lower-risk myelodysplastic syndromes: a phase 2 clinical trial. Nat Commun. 2024 Nov 13;15(1):9840. doi: 10.1038/s41467-024-54290-2. PMID 39537648
- See also: MD Anderson Cancer Center — http://www.mdanderson.org